CLINICAL TRIAL: NCT06262633
Title: A Multi-centre Trial on Targeted Microwave Ablation (TMA) for Localized Prostate Cancer Using Organ Based Tracking (OBT) Navigation
Brief Title: A Multi-centre Trial on Targeted Microwave Ablation (TMA) for Localized Prostate Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, CHIU Ka Fung Peter, Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRE-2023.079
Record Dates: First submitted 2024-01-21; First posted 2024-02-16 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Targeted Microwave Ablation (TMA) (Experimental): Targeted Microwave Ablation (TMA) for localized prostate cancer using organ based tracking (OBT) navigation
  Interventions: Device: Targeted Microwave Ablation (TMA) for localized prostate cancer using organ based tracking (OBT) navigation

INTERVENTIONS:
Device: Targeted Microwave Ablation (TMA) for localized prostate cancer using organ based tracking (OBT) navigation — Targeted microwave ablation (TMA) is a novel treatment developed for focal treatment of prostate cancer, and it is applied with precise navigation guidance under the organ-based tracking (OBT) mechanism.

SUMMARY:
This study is to investigate the efficacy of Targeted Microwave Ablation (TMA) under MRI-Ultrasound fusion and organ-based tracking (OBT) navigation in localized prostate cancer (PCa) in a multi-centre trial.

DETAILED DESCRIPTION:
This is a prospective multi-centre trial in 5 hospitals in 3 countries to investigate the efficacy and complications of targeted Microwave Ablation as a minimally invasive focal therapy for prostate cancer. Men aged 50-75 with PSA < 20ng/mL and clinically significant prostate cancer with 1-2 MRI lesions ≤15mm and ISUP grade group ≤3 will be recruited. Transperineal targeted Microwave Ablation of the prostate tumor(s) will be done with repeated ablations by a single microwave needle guided by MRI-Ultrasound fusion and organ-based tracking navigation. The primary outcome is any clinically significant prostate cancer detected on biopsy of treated area(s) per patient at 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Men aged between 45 - 75 years
2. Life expectancy > 10 years upon recruitment
3. Able to understand the trial and can provide informed and written consent, dated and signed before the enrollment and before any exam required by the trial
4. Localized low or intermediate risk prostate cancer diagnosed on MRI-Ultrasound fusion targeted biopsy
5. Organ-confined prostate cancer on MRI
6. PSA < 20 ng/mL
7. 1-2 MRI visible lesion present and size ≤15mm, with targeted biopsy showing:

   * ISUP grade group 2 or 3, or
   * ISUP grade group 1 with tumor size ≥10mm

Exclusion Criteria:

1. Patients not fit for general or spinal anaesthesia
2. Patients unfit for MRI exam or MR gadolinium contrast (e.g. estimated glomerular filtration rate (eGFR) of <50 ml/min)
3. Patients with coagulopathy that cannot be corrected
4. Patients on anticoagulants or antiplatelets that cannot be stopped (Low dose Aspirin, e.g. 80-100mg, is acceptable and no need to stop before or during TMA treatment)
5. Patients with previous treatment of prostate cancer
6. Patients with prior pelvic radiotherapy for prostate cancer or other cancer
7. Patients with maximal length of target lesion >15mm
8. Patients with MRI-visible or invisible lesion within 10mm from rectum or 10mm from sphincter on MRI
9. . Patients with >2 areas (MRI-visible or invisible) of prostate cancer
10. Patients with Gleason score 4+4 or any Gleason pattern 5 cancer
11. Patients with systematic cores showing any Gleason 4 pattern PCa which are not adjacent to the target lesions (1 core of pure Gleason 3 pattern PCa on systematic cores in contralateral lobe is acceptable)
12. Patients with definite cT3 or above disease on imaging (prostate capsular contact without definite extra-capsular extension is acceptable)
13. Patients with bladder pathology including bladder stone and bladder cancer
14. Patients with known urethral stricture
15. Patient with a suspected COVID-19 disease or an active SARS-CoV-2 infection.

Ages: 45 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 103 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
The oncological control of prostate cancer | At 6 months after treatment
  Any cancer detected on biopsy of each ablated area

SECONDARY OUTCOMES:
Cancer detection on biopsy of each ablated MRI visible lesion | At 6 months after treatment
  Cancer detection on biopsy of each ablated MRI visible lesion
Cancer detection on biopsy of each ablated MRI invisible lesion | At 6 months after treatment
  Cancer detection on biopsy of each ablated MRI invisible lesion
Gleason 4 or 5 cancer detected on biopsy of ablated area | At 6 months after treatment
  The higher the Gleason score, the higher grade the prostate cancer
Out-of-field recurrence: Any cancer outside treated area on systematic biopsy | At 6 months after treatment
  Out-of-field recurrence: Any cancer outside treated area on systematic biopsy
Common Terminology Criteria for Adverse Events (CTCAE) v5.0 | At 3 Month, 6 Month and 1 year
  Complications of treatment using Common Terminology Criteria for Adverse Events (CTCAE) v5.0
PSA change | At baseline, 3 Month and 6 Month and 12 Month
  PSA change after treatment
Urinary Symptoms after treatment | At baseline, 3 Month, 6 Month and 12 Month
  Urinary symptoms measured by IPSS score, score ranging from 0-35 (the higher the worse)
Sexual side effects after treatment | At baseline, 3 Month, 6 Month and 12 Month
  Sexual side effects, up to 1 year, measured by IIEF-5 score (ranging from 1-25), the lower the worse
Continence side effects after treatment | At baseline, 3 Month, 6 Month and 12 Month
  Continence side effects, up to 1 year, measured by EPIC-26 questionnaire, the higher score the lower score the worse
Common Terminology Criteria for Adverse Events (CTCAE) rectal toxicity | At baseline, 3 Month, 6 Month and 12 Month
  Rectal toxicity of treatment using Common Terminology Criteria for Adverse Events
Quality of life measured by ED-5Q-5Lquestionnaire | At baseline, 3 Month, 6 Month and 12 Month
  Quality of life measured by ED-5Q-5L questionnaire, the higher the score the better in quality of life
Quality of life in patients with prostate cancer measured by EPIC-26 | At baseline, 3 Month, 6 Month and 12 Month
  Quality of life in patients with prostate cancer measured by EPIC-26 range 0-100, the higher score the better the quality of life
Quality of life measured by QLQ-C30, | At baseline, 3 Month, 6 Month and 12 Month
  Quality of life measured by QLQ-C30, score 0-100, the higher the score the better in quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Peter Ka-Fung CHIU, PhD,MBChB, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Peter Ka-Fung CHIU, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Culp MB, Soerjomataram I, Efstathiou JA, Bray F, Jemal A. Recent Global Patterns in Prostate Cancer Incidence and Mortality Rates. Eur Urol. 2020 Jan;77(1):38-52. doi: 10.1016/j.eururo.2019.08.005. Epub 2019 Sep 5. PMID 31493960
- [Background] Rawla P. Epidemiology of Prostate Cancer. World J Oncol. 2019 Apr;10(2):63-89. doi: 10.14740/wjon1191. Epub 2019 Apr 20. PMID 31068988
- [Background] Stabile A, Orczyk C, Hosking-Jervis F, Giganti F, Arya M, Hindley RG, Dickinson L, Allen C, Punwani S, Jameson C, Freeman A, McCartan N, Montorsi F, Briganti A, Ahmed HU, Emberton M, Moore CM. Medium-term oncological outcomes in a large cohort of men treated with either focal or hemi-ablation using high-intensity focused ultrasonography for primary localized prostate cancer. BJU Int. 2019 Sep;124(3):431-440. doi: 10.1111/bju.14710. Epub 2019 Mar 18. PMID 30753756
- [Background] Durand M, Barret E, Galiano M, Rozet F, Sanchez-Salas R, Ahallal Y, Macek P, Gaya JM, Cerruti J, Devilliers H, Loeffler J, Amiel J, Vallancien G, Cathelineau X. Focal cryoablation: a treatment option for unilateral low-risk prostate cancer. BJU Int. 2014 Jan;113(1):56-64. doi: 10.1111/bju.12370. Epub 2013 Oct 31. PMID 24053685
- [Background] Shah TT, Peters M, Eldred-Evans D, Miah S, Yap T, Faure-Walker NA, Hosking-Jervis F, Thomas B, Dudderidge T, Hindley RG, McCracken S, Greene D, Nigam R, Valerio M, Minhas S, Winkler M, Arya M, Ahmed HU. Early-Medium-Term Outcomes of Primary Focal Cryotherapy to Treat Nonmetastatic Clinically Significant Prostate Cancer from a Prospective Multicentre Registry. Eur Urol. 2019 Jul;76(1):98-105. doi: 10.1016/j.eururo.2018.12.030. Epub 2019 Jan 9. PMID 30638633
- [Background] Barry Delongchamps N, Schull A, Anract J, Abecassis JP, Zerbib M, Sibony M, Jilet L, Abdoul H, Goffin V, Peyromaure M. Feasibility and safety of targeted focal microwave ablation of the index tumor in patients with low to intermediate risk prostate cancer: Results of the FOSTINE trial. PLoS One. 2021 Jul 14;16(7):e0252040. doi: 10.1371/journal.pone.0252040. eCollection 2021. PMID 34260598
- [Background] Chiu PK, Chan CH, Yee CH, Lau SY, Teoh JY, Wong HF, Lo KL, Yuen TY, Hung HY, Cho CC, Ng CF. Transperineal Targeted Microwave Ablation (TMA) of localized prostate cancer guided by MRI-Ultrasound fusion and organ-based tracking: a pilot study. Prostate Cancer Prostatic Dis. 2023 Dec;26(4):736-742. doi: 10.1038/s41391-022-00577-8. Epub 2022 Jul 14. PMID 35835844
- [Background] Turkbey B, Rosenkrantz AB, Haider MA, Padhani AR, Villeirs G, Macura KJ, Tempany CM, Choyke PL, Cornud F, Margolis DJ, Thoeny HC, Verma S, Barentsz J, Weinreb JC. Prostate Imaging Reporting and Data System Version 2.1: 2019 Update of Prostate Imaging Reporting and Data System Version 2. Eur Urol. 2019 Sep;76(3):340-351. doi: 10.1016/j.eururo.2019.02.033. Epub 2019 Mar 18. PMID 30898406